

# Protocol for observational studies based on existing data

| Document Number: | c02329987-02 |
|---|---|
| BI Study Number: | 1222.53 |
| BI Investigational Product(s): | Olodaterol |
| Title: | Drug Utilisation Study for Olodaterol |
| Protocol version identifier: | Version 2.0 |
| Date of last version of protocol: | 13 Feb 2014 |
| PASS: | Yes |
| EU PASS register number: | Study not registered |
| Active substance: | Olodaterol |
| Medicinal product: | Striverdi, Respimat |
| Product reference: | BI 1744 |
| Procedure number: | Not applicable |
| Marketing authorisation holder(s): | Boehringer Ingelheim GmbH |
| Joint PASS: | No |
| Date: | 14 Oct 2014 |

Proprietary confidential information

© 2014 Boehringer Ingelheim International GmbH or one or more of its affiliated companies. All rights reserved.

This document may not - in full or in part - be passed on, reproduced, published or otherwise used without prior written permission

Proprietary confidential information © 2014 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# **Additional Information**

| | I |
|---|---|
| Research question and objectives: | This study aims to characterise the use of single-agent olodaterol and single-agent indacaterol, the only marketed long-acting beta2-agonist (LABAs) authorised for chronic obstructive pulmonary disease (COPD), but not for asthma, in clinical practice. Study objectives are as follows: Primary objectives: |
| | <ul> <li>Quantify the frequency of off-label use of olodaterol among new users of these medications (i.e., the proportion of new users who do not have COPD)</li> <li>Describe the baseline characteristics of new users of olodaterol</li> </ul> |
| | Secondary objective: |
| | <ul> <li>Quantify the frequency of off-label use of indacaterol (a LABA approved for COPD but not for asthma) among new users of these medications (i.e., the proportion of new users who do not have COPD), in order to put into perspective the results for olodaterol initiators</li> <li>Describe the baseline characteristics of new users of indacaterol</li> </ul> |
| Country(-ies) of study: | The Netherlands, Denmark, and Sweden |
| Author: | |
| Marketing authorisation holder(s): | |
| MAH contact person: | |
| EU-QPPV: | |
| Signature of EU-QPPV: | The signature of the EU-QPPV is provided electronically |

Proprietary confidential information © 2014 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# 1. TABLE OF CONTENTS

| TITI | LE PAG | E | 1 |
|---|---|---|---|
| 1. | TABL | E OF CONTENTS | 3 |
| 2. | LIST ( | OF ABBREVIATIONS | 6 |
| 3. | RESPO | ONSIBLE PARTIES | 8 |
| 4. | ABST | RACT | 9 |
| 5. | AMEN | IDMENTS AND UPDATES | 11 |
| 6. | MILES | STONES | 12 |
| 7. | RATIO | ONALE AND BACKGROUND | 13 |
| 8. | RESEA | ARCH QUESTION AND OBJECTIVES | 14 |
| 9. | RESEA | ARCH METHODS | 15 |
| 9.1 | STU | JDY DESIGN | 15 |
| 9.2 | SET | TING | 15 |
| 9 | 9.2.1 | Source population | 18 |
| Ģ | 9.2.2 | Study period | 18 |
| 9 | 9.2.3 | Study groups | 18 |
| | 9.2.3.1 | Inclusion criteria | 19 |
| | 9.2.3.2 | 2 Exclusion criteria | 19 |
| 9.3 | VA | RIABLES | |
| Ģ | 9.3.1 | Exposures | |
| Ģ | 9.3.2 | Indication and potential off-label prescribing | |
| | 9.3.2.1 | | |
| | 9.3.2.2 | | |
| | 9.3.2.3 | 1 1 | |
| | | 1 Classification of patients | |
| ç | 9.3.3 | Characterisation of new users of olodaterol and indacaterol | |
| | 9.3.3.1 | | |
| | 9.3.3.2 | 1 J J | |
| | 9.3.3.3 | , | |
| | 9.3.3.4 | 3 | |
| | 9.3.3.5 | 3 | |
| | 9.3.3.6 | | |
| - | 9.3.3.7 | | |
| 9 | 9.3.4 | Outcomes | 28 |

| Proprietary confid | lential information © 2014 Boehringer Ingelheim International GmbH or one or more of its affiliated comp | anies |
|---|---|---|
| 9.3.4. | Primary outcome | 28 |
| 9.3.4.2 | 2 Secondary outcomes | 29 |
| 9.3.4.2<br>new u | The secondary outcome is the prevalence of off-label prescribing are sers of indacaterol | _ |
| 9.3.5 | Covariates | 29 |
| 9.4 DA | TA SOURCES | 29 |
| 9.4.1 | PHARMO Database Network | 29 |
| 9.4.1. | Database characteristics | 29 |
| 9.4.2 | Denmark | 30 |
| 9.4.3 | Sweden | 30 |
| 9.4.4 | Summary of study databases | . 31 |
| 9.5 STU | JDY SIZE | 34 |
| 9.6 DA | TA MANAGEMENT | 35 |
| 9.7 DA | TA ANALYSIS | 36 |
| 9.7.1 | Main analysis | 36 |
| 9.7.2 | Indication and potential off-label prescribing | 36 |
| 9.7.3 | Number of users and patterns of use | 36 |
| 9.7.4 | Characterisation of new users at the index date | . 36 |
| 9.8 QU | ALITY CONTROL | . 38 |
| 9.9 LIM | IITATIONS OF THE RESEARCH METHODS | . 38 |
| 9.10 OT | HER ASPECTS | . 39 |
| 9.10.1 | Bias | . 39 |
| 10. PROT | ECTION OF HUMAN SUBJECTS | 40 |
| | AGEMENT AND REPORTING OF ADVERSE EVENTS/ADVERSE TIONS | 41 |

12. PLANS FOR DISSEMINATING AND COMMUNICATING STUDY RESULTS 42

13. REFERENCES 43

EVALUATION OF COPD SEVERITY IN AUTOMATED HEALTH

ANNEX 4. CODES FOR COMORBIDITIES AND OTHER MEDICATIONS...... 58

13.1

13.2

ANNEX 1.

ANNEX 2.

ANNEX 3.

| Boehringer Ingelheim | |
|-----------------------------------------------------------|--------------|
| Protocol for observational studies based on existing data | S |
| BI Study Number 1222.53 | c02329987-02 |

| Proprietary confidential information © 2014 Boehringer Ingelheim International GmbH or one or m | ore of its affiliated companies |
|---|---|
|---|---|

| ANNEX 5. | DETAILS ON | EACH DA | TABASE | FROM | THE FE | ASIBILIT <b>`</b> | Y REPORT |
|---|---|---|---|---|---|---|---|
| (1 NO | <b>VEMBER 2013)</b> | | | | | | 64 |

Proprietary confidential information © 2014 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## 2. LIST OF ABBREVIATIONS

AMI Acute Myocardial Infarction

ATC Anatomical Therapeutic Chemical

BI Boehringer Ingelheim

BMI Body Mass Index

CAT COPD Assessment Test

COPD Chronic Obstructive Pulmonary Disease

DAMD Danish General Practice Database

DDD Defined Daily Dose

EMA European Medicines Agency

ENCePP European Network of Centres for Pharmacoepidemiology and

Pharmacovigilance

FEV<sub>1</sub> Forced Expiratory Volume in 1 Second

GOLD Global Initiative for Chronic Obstructive Lung Disease

GP General Practitioner or General Practice
ICD International Classification of Diseases

ICD-10 International Statistical Classification of Diseases and Related Health

Problems, 10th Revision

ICD-10-CM International Statistical Classification of Diseases and Related Health

Problems, 10th Revision, Clinical Modification

ICD-9 International Classification of Diseases, 9th Revision

ICD-9-CM International Classification of Diseases, 9th Revision, Clinical Modification

ICPC International Classification of Primary Care

ICS Inhaled Glucocorticosteroid LABA Long-Acting Beta2-Agonist

LAMA Long-Acting Muscarinic Antagonist

mMRC Modified British Medical Research Council Questionnaire

NCSP Nordic Medico-Statistical Committee Classification of Surgical Procedures

NPR National Patient Register (Sweden)
PASS Post-Authorisation Safety Study

PHARMO Institute for Drug Outcomes Research (the Netherlands); also short for the

PHARMO Database Network

PHARMO-GP a data subset of PHARMO Database Network with information from GPs

PPV Positive Predictive Value

# Boehringer Ingelheim Protocol for observational studies based on existing data BI Study Number 1222.53

**** 

c02329987-02

Proprietary confidential information © 2014 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

PRO Patient-Reported Outcome

SABA Short-Acting Beta2-Agonist

SAMA Short-Acting Muscarinic Antagonist

SD Standard Deviation

WHO World Health Organization

Proprietary confidential information © 2014 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## 3. RESPONSIBLE PARTIES

The following individual is the author of this protocol:

The following individuals have collaborated with the author on protocol development.

, RTI Health Solutions RTI Health Solutions

## The following institutions will implement the study:

PHARMO Institute, the Netherlands Denmark – To be determined Karolinska Institutet, Sweden

Note: Investigators at these institutions will be named after they have reviewed the protocol and agreed to participate.

Proprietary confidential information © 2014 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# 4. ABSTRACT

| Name of company: | | | |
|---|---|---|---|
| Boehringer Ingelheim GmbH | | | |
| Name of finished medicina<br>Striverdi, Respimat | al product: | | |
| Name of active ingredient<br>Olodaterol | • | | |
| Protocol date: | Study number: | Version/Revision: | Version/Revision date: |
| 13 Feb 2014 | 1222.53 | 2.0 | 14 Oct 2014 |
| Title of study: | Drug Utilisation Stud | ly for Olodaterol | |
| Rationale and background: | Boehringer Ingelheim GmbH (BI) developed olodaterol, an inhaled long-acting beta2-agonist (LABA), for the indication of chronic obstructive pulmonary disease (COPD). LABAs are used in COPD to relieve bronchial constriction and, consequently, to improve symptoms. Because the use of LABAs has been associated with increased morbidity and mortality in patients with asthma, within the "Decentralised Procedure for Striverdi Respimat" the health authorities of the European Union/European Economic Area Member States requested the conduct of a post-approval drug utilisation study to assess potential off-label use of olodaterol in asthma and to characterise the use of olodaterol in clinical practice. | | |
| Research question and objectives: | <ul> <li>This study aims to characterise the use of single-agent olodaterol and single-agent indacaterol, the only marketed LABAs authorised for COPD, but not for asthma, in clinical practice. Study objectives are as follows:</li> <li>Primary objectives:</li> <li>Quantify the frequency of off-label use of olodaterol among new users of these medications (i.e., the proportion of new users who do not have COPD)</li> <li>Describe the baseline characteristics of new users of olodaterol</li> <li>Secondary objective:</li> <li>Quantify the frequency of off-label use of indacaterol (a LABA approved for COPD but not for asthma) among new users of these medications (i.e., the proportion of new users who do not have COPD), in order to put into perspective the results for olodaterol initiators</li> </ul> | | |
| Study design: | Describe the baseline characteristics of new users of indacaterol This is a cross-sectional study using information collected in health care databases among new users of olodaterol or indacaterol in the Netherlands, Denmark, and Sweden. | | |

Proprietary confidential information © 2014 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| Population: | The source population is all subjects enrolled in the selected study databases at the date olodaterol and indacaterol are available in each database's country. The study groups are those subjects from the source population who receive a first dispensing for single-agent formulations of olodaterol for the primary objective or indacaterol for the secondary objective and have at least 12 months of continuous enrolment in the study databases. |
|---|---|
| Variables: | Indication and potential off-label use of olodaterol and indacaterol; characterisation of new users of olodaterol and indacaterol by demographic variables, medical history, and use of other medications. |
| Data sources: | The study is planned to be conducted in the following databases: the PHARMO Database Network in the Netherlands, the National Registers in Denmark, and the National Registers in Sweden A description of each database is provided in Section 9.4; further details from the feasibility report are provided in ANNEX 5. The study will be conducted by using data on drug prescriptions and disease occurrence routinely collected on an ongoing basis for large population-based automated health care databases in the Netherlands, Denmark, and Sweden. |
| Study size: | Actual counts of numbers of patients using olodaterol in European countries are not yet available since it is not yet marketed in Europe. |
| Data analysis: | Number and proportion of new users by indication and potential off-<br>label use. Number and proportion of new users according to medical<br>history and use of comedications |
| Milestones: | Start of data collection (contingent on approval, reimbursement, and uptake of olodaterol): • Denmark: Q1 2015 • The Netherlands: Q4 2015 • Sweden: Q4 2015 End of data collection: Q1 2018 Interim reports of study results: Q3 2017 Final report of study results: Q3 2018 |

Proprietary confidential information © 2014 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# 5. AMENDMENTS AND UPDATES

Version 2.0 includes clarification to the milestone table and revision of the primary and secondary study objectives in the context of regulatory review of the protocol.

| Number | Date | Section of<br>Study<br>Protocol | Amendment or<br>Update | Reason |
|---|---|---|---|---|
| 1 | 30 Sep<br>2014 | 6 | Update of milestones | Delay in finalization of protocol to respond to regulatory authority review |
| 2 | 30 Sep<br>2014 | 8 | Research objectives | Modified in response to regulatory authority review |
| 3 | 30 Sep<br>2014 | 9.3.4 | Clarification of primary outcomes | Modified in response to regulatory authority review |

Proprietary confidential information © 2014 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## 6. MILESTONES

| Milestone | Planned Date <sup>1</sup> |
|---|---|
| Start of data collection (expected availability of data on earliest exposure group entry)2: | Denmark: Q1 2015<br>The Netherlands: Q4 2015<br>Sweden: Q4 2015 |
| End of data collection (latest possible exposure group entry): | Denmark: Q1 2018 The Netherlands: Q1 2018 Sweden: Q1 2018 |
| Study progress report(s): | TBD |
| Interim report(s) of cumulative study results: | Q3 2017 |
| Registration in the EU PAS register: | After regulatory endorsement of the protocol |
| Final report of study results from all databases: | Q3 2018 |

TBD = to be determined. Contact with database custodians is pending.

- Preliminary; dependent on market uptake of olodaterol and contracts with MAH and research partners.
- Considering launch dates and approximately 1-year lag time in database. Launch dates are March 2014 in Denmark, February 2014 in the Netherlands, and August 2014 in Sweden.

Proprietary confidential information © 2014 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# 7. RATIONALE AND BACKGROUND

Chronic obstructive pulmonary disease (COPD) is a serious, chronic disease that affects millions of people worldwide. [P13-02399] COPD typically involves persistent limitation of airflow, a progressive course, and chronically enhanced inflammatory response of the airways to airborne particulates and gases. [P13-02399]

Worldwide, the estimated number of patients with COPD is 63.6 million. [R09-2531] In 2004, the World Health Organization estimated that the European region had approximately 11.3 million patients with prevalent, symptomatic COPD. [R09-2531] A systematic review and meta-analysis of 67 studies conducted in 28 countries between 1990 and 2004 showed that the prevalence of COPD is higher in subjects over 40 years of age than those under 40. The pooled prevalences were 3.1% in subjects under 40 years of age and 9.9% in those 40 years old or older, 8.2% for ages 40-64, and 14.2% for ages 65 years or older. [R06-4117] The health, social, and economic burdens of COPD are predicted to increase in the next several decades because of continuing exposure to tobacco smoke and other risk factors and because of the increasing age of the general populations in many countries. [P13-02399]

Inhaled long-acting beta2-agonist (LABA) drugs are used in COPD and in asthma. At present, the approved indication for the three major LABAs in COPD, formoterol, salmeterol, and indacaterol, is maintenance or long-term use. Formoterol and salmeterol are also approved for use in asthma; for this condition, simultaneous use with corticosteroids is strongly recommended. Within the Decentralised Procedure for Striverdi Respimat, the health authorities of the European Union/European Economic Area Member States requested the conduct of a post-approval drug utilisation study to assess the potential off-label use of olodaterol in asthma patients and to characterise the use of olodaterol in clinical practice.

This protocol is a core protocol describing the study design, methods, and analysis for implementing the study in three European health care databases in the Netherlands, Denmark, and Sweden. This core protocol will need to be adapted to the specifics of each database regarding the type and availability of the recorded information and the coding systems used to record diagnoses and medications.

Proprietary confidential information © 2014 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# 8. RESEARCH QUESTION AND OBJECTIVES

This study aims to assess the use of single-agent olodaterol in clinical practice. The single agent indacaterol, the only marketed LABA authorised in clinical practice for COPD but not for asthma, will also be assessed. Study objectives are as follows:

## Primary objectives:

- Quantify the frequency of off-label use of olodaterol among new users of these medications (i.e., the proportion of new users who do not have COPD)
- Describe the baseline characteristics of new users of olodaterol

## Secondary objectives:

- Quantify the frequency of off-label use of indacaterol (a LABA approved for COPD but not for asthma) among new users of these medications (i.e., the proportion of new users who do not have COPD), in order to put into perspective the results for olodaterol initiators
- Describe the baseline characteristics of new users of indacaterol

Proprietary confidential information © 2014 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## 9. RESEARCH METHODS

#### 9.1 STUDY DESIGN

This is a cross-sectional study using information collected in health care database(s) among new users of olodaterol or indacaterol in the Netherlands, Denmark, and Sweden. The study period will be 3 consecutive years, with annual cross-sectional descriptions of new users of olodaterol and indacaterol. Evaluation of off-label use and characterisation of new users will be conducted at the **index date**, defined as the date an eligible patient receives the first dispensing of olodaterol or indacaterol.

#### 9.2 SETTING

The study is planned to be conducted in the following databases: the PHARMO Database Network in the Netherlands, the National Registers in Denmark, and the National Registers in Sweden. The type of data available in each database is summarised in Table 1. A detailed description of each study database is provided in Sections 9.4, 9.4.2 and 9.4.3.

Proprietary confidential information © 2014 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Table 1 Selected characteristics of the study databases

| Type of Data | PHARMO,<br>the Netherlands | National<br>Registers,<br>Denmark | National<br>Registers,<br>Sweden |
|---|---|---|---|
| Hospital inpatient discharge diagnoses | Yes | Yes | Yes |
| Hospital inpatient procedures | Yes | Yes | Yes |
| Hospital/clinics outpatient diagnoses | No | Yes | Yes |
| General practitioner diagnoses | Yes, in data subset<br>PHARMO-GP <sup>1</sup> | Yes, for selected<br>general practices<br>in the Danish<br>General Practice<br>Database <sup>2</sup> | Yes, for general practices from the counties of Stockholm and Göteborg <sup>3</sup> |
| Pharmacy-dispensed medications | Yes | Yes | Yes |
| Prescribed medications | Yes in data subset<br>PHARMO-GP <sup>1</sup> | Yes <sup>2</sup> | Yes <sup>3</sup> |

#### GP = General Practitioner.

- 1 PHARMO-GP includes approximately 440,000 subjects.
- 2 The Danish General Practice Database includes approximately 1 million subjects.
- 3 Population from the counties of Stockholm and Göteborg is about 25% of the total Swedish population

In each country, new users of olodaterol and indacaterol will be identified in the prescription databases, which record information on the medications dispensed in the pharmacies (Figure 1). New users will be characterised in terms of past medical history and use of medications. Past medical history will be evaluated by linkage via unique patient-specific identifiers using the hospitalisation databases, which provide information on hospital and outpatient discharge diagnoses and procedures. Use of medications will be evaluated using the prescription databases. Off-label prescribing will be evaluated for those new users for whom general practitioner diagnoses are available because information from general practitioners is considered the most appropriate for evaluating the indication and potential off-label use of medications.

Proprietary confidential information © 2014 Boehringer Ingelheim International GmbH or one or more of its affiliated companies



Figure 1 Overall study design

The coding of diagnoses and procedures varies across databases (Table 2). In PHARMO, diagnoses are coded using the *International Classification of Diseases, 9th Revision* (ICD-9); whereas in Denmark and Sweden, diagnoses are coded using the *International Statistical Classification of Diseases and Related Health Problems, 10th Revision* (ICD-10). In PHARMO, procedures are coded using ICD-9 codes; in Denmark, using ICD-10 codes; and in Sweden, using the 2012 Nordic Medico-Statistical Committee's Classification of Surgical Procedures, version 1.16.[R14-0443] The Anatomical Therapeutic Chemical (ATC) classification is used in all three databases to code dispensed medications.

Proprietary confidential information © 2014 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Table 2 Types of diagnosis, procedures, and medication codes in the study databases

| Type of Code | PHARMO,<br>The Netherlands | National Registers,<br>Denmark | National<br>Registers, Sweden |
|---|---|---|---|
| Diagnoses | Hospital: ICD-9 | ICD-10 | ICD-10 |
| | Primary health care: ICPC <sup>1</sup> | Primary health care: ICPC <sup>1</sup> | |
| Procedures | ICD-9 | ICD-10 | NCSP 1.16, 2012 |
| Medications | ATC | ATC | ATC |

ATC = Anatomical Therapeutic Chemical; GP = General Practitioner; ICD-9 = International Classification of Diseases, 9th Revision; ICD-10 = International Statistical Classification of Diseases and Related Health Problems, 10th Revision; ICPC = International Classification of Primary Care; NCSP = Nordic Medico-Statistical Committee's Classification of Surgical Procedures.

### 9.2.1 Source population

The study source population includes all subjects enrolled in the selected study databases at the date olodaterol and indacaterol are available in each database's country.

# 9.2.2 Study period

The start of the study period is at the index date, defined as the dates of the first recorded dispensings of olodaterol and indacaterol in each database. New users of olodaterol and indacaterol will be identified in each of 3 consecutive years, with annual cross-sectional evaluations of off-label use and of characteristics of users.

#### 9.2.3 Study groups

Study groups are those subjects from the source population who (1) receive a first dispensing for single-agent formulations of olodaterol or indacaterol and (2) have at least 12 months of continuous enrolment in the study databases preceding the index date. Two study groups will be created: (1) a group of new users of olodaterol and (2) a group of new users of indacaterol.

New users of olodaterol are defined as patients who, with at least 12 months of continuous enrolment before the index date, have their first record of a dispensing for olodaterol. Similarly, new users of indacaterol have their first record of a dispensing for indacaterol in the database (after at least 12 months of continuous enrolment). Patients who receive a dispensing for olodaterol or indacaterol before they meet the criteria of 12 months of continuous enrolment in the database are not eligible to enter the corresponding study groups (olodaterol or indacaterol).

Each group of new users of olodaterol and new users of indacaterol will be divided into two subgroups: (1) LABA naïve in the short term (3 months) and (2) switchers from another LABA. Patients who are LABA naïve in the short term are defined as any new users of olodaterol or indacaterol who did not receive any dispensing for LABAs within 3 months

<sup>1</sup> Available for PHARMO-GP, a data subset of PHARMO with information from GPs.

Proprietary confidential information © 2014 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

before the index date. Switchers are defined as any new user of olodaterol or indacaterol who received a dispensing for a different LABA within the 3 months before the index date. Within the olodaterol group and within the indacaterol group, LABA-naïve patients and switchers will be described and compared.

#### 9.2.3.1 Inclusion criteria

To be included in a study group, patients must have at least 12 consecutive months of enrolment in the database before the index date. This will allow evaluation of the medical history and prior use of medications of included patients.

#### 9.2.3.2 Exclusion criteria

Because the study aims to assess the use of olodaterol and indacaterol in regular clinical practice, no exclusions regarding age, sex, or comorbidity will be defined. However, individuals with missing or implausible values for age or sex will be excluded.

#### 9.3 VARIABLES

# 9.3.1 Exposures

New users of olodaterol and indacaterol will be identified at the first record of a dispensing for the relevant medication code specific to each database. New users are defined in Section 9.2.3. The ATC code for indacaterol is R03AC18, classified as a selective beta2-adrenoreceptor agonist in the category of inhalant adrenergics. Indacaterol is available as inhalation powder with a defined daily dose (DDD) of 0.15 mg. The ATC code for olodaterol is R03AC19.

## 9.3.2 Indication and potential off-label prescribing

The indication for the prescribing of medications are not recorded in the study databases; therefore, the indication of treatment and potential off-label use of olodaterol and indacaterol will be inferred from the diagnoses codes recorded before the index date or at the index date and complemented by the clinical review of the computerised information. The indication and potential off-label use will be evaluated in the subset of new users whose information is linked to the general practice (primary care) registers that include diagnoses recorded by general practitioners. Information from general practitioners is considered the most appropriate for assessing the indication and potential off-label use of medications. Primary care data are available in the following study databases:

- PHARMO-GP covering about 440,000 population
- Danish General Practice Database covering about 1 million population
- Swedish General Practice Database in the counties of Stockholm and Göteborg

Potential off-label use will be evaluated separately by the following age groups:

- 0 to 17 years
- 18 to 29 years
- 30 to 39 years

Proprietary confidential information © 2014 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

- 40 to 49 years
- 50 to 59 years
- 60 to 69 years
- 70 to 79 years
- 80 years and older

## 9.3.2.1 On-label prescribing: indication of COPD

The indication of COPD is defined as any patient with a diagnosis of COPD, chronic bronchitis, or emphysema recorded in the database at any time before the index date or at the index date. Because COPD can occur in association with asthma, patients with a recorded diagnosis for both COPD and asthma will be considered on-label. [R14-0350] [R07-2620] [R08-1492].

For this study, classification of COPD status will be based on general practice diagnoses and hospital outpatient and inpatient discharge diagnoses. No validation data are available for COPD diagnoses recorded in PHARMO. In general, in Denmark and Sweden, validation has been performed for COPD diagnoses ascertained via hospital (inpatient and outpatient) diagnoses. ICD diagnoses codes for COPD have shown a good positive predictive value (PPV). In the Danish National Registers, the PPV for the hospital discharge diagnosis of COPD (ICD-10 code J44) was 92%. [R14-0359] In Sweden, a COPD validation study showed that the COPD diagnosis (ICD-9: 491-492, 496; ICD-10: J41-J44) recorded in the National Inpatient Registry was considered as proven in 21.7% of cases, probable in 35.5%, possible in 34.0%, uncertain in 2.1%, and unlikely in 7.0%. [R14-0456] The proportion of patients with asthma misclassified as having COPD was 2.1%, and the overall degree of misclassification was less than 10%. The registry was considered of acceptable validity for epidemiological research of COPD.

The ICD-10 and ICD-9 codes to identify the diagnosis of COPD are detailed in Table 3. Diagnosis codes include COPD, chronic bronchitis, and emphysema.

Proprietary confidential information © 2014 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Table 3 ICD-10 and ICD-9 diagnoses and codes to identify patients with COPD

| ICD-10 Code Description | ICD-10 Code | ICD-9 Code |
|---------------------------------------------|-------------|------------|
| Chronic bronchitis | J41-J42 | 491 |
| Emphysema | J43 | 492 |
| Other COPD | J44 | 496 |
| COPD with acute lower respiratory infection | J44.0 | _ |
| COPD with acute exacerbation, unspecified | J44.1 | _ |
| Other specified COPD | J44.8 | _ |
| COPD, unspecified | J44.9 | _ |

COPD = Chronic Obstructive Pulmonary Disease; ICD-9 = International Classification of Diseases, 9th Revision; ICD-10 = International Statistical Classification of Diseases and Related Health Problems, 10th Revision.

#### 9.3.2.2 Off-label prescribing

Patients without a recorded diagnosis of COPD at any time before the index date or patients with a recorded diagnosis of asthma in the absence of a diagnosis for COPD will be considered off-label users. The off-label prescribing of olodaterol and indacaterol for the treatment of asthma is of special interest because this class of medication is often used in asthma but olodaterol and indacaterol have not been developed or approved for asthma.

Few studies have examined the validity of ICD codes for identifying patients with asthma. In a validation study conducted in Sweden, the PPV for the diagnosis of asthma (ICD-10 J45) associated with visits to outpatient specialty clinics and inpatient stays and recorded in the National Patient Registry among patients 18 to 45 years of age treated with asthma medications was 89% (95% confidence interval, 83%-93%). [R14-0349] The proportion of subjects misclassified as COPD was 1.6%. In another study conducted in the RAMQ Medical Services database of the province of Quebec in Canada, the PPV for having one or more recorded diagnoses of asthma (ICD-9 493) over a 1-year period in patients aged 16 to 44 years was 75% when the diagnosis was recorded by respiratory physicians and 67% when it was recorded by family physicians. The PPV increased to 77% for respiratory physicians and to 78% for family physicians when two or more recorded diagnoses of asthma were required. [R14-0352] Another study conducted in children under 4 years of age using data from the Rochester Epidemiology Project database showed that the overall agreement of ICD code 493 and information from the medical chart was 81.6%. [R14-0351]

The ICD-10 and ICD-9 codes to identify patients with asthma are detailed in Table 4.

Proprietary confidential information © 2014 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Table 4 ICD-10 and ICD-9 diagnoses and codes to identify patients with asthma

| ICD-10 Code Description | ICD-10 Code | ICD-9 Code |
|-------------------------------|-------------|--------------------|
| Asthma | J45 | 493 |
| Predominantly allergic asthma | J45.0 | 493.0 <sup>1</sup> |
| Non-allergic asthma | J45.1 | 493.11 |
| Mixed asthma | J45.8 | _ |
| Asthma, unspecified | J45.9 | 493.9 <sup>1</sup> |
| Chronic obstructive asthma | | 493.2 <sup>1</sup> |
| Other forms of asthma | | 493.8 |
| Status asthmaticus | J46 | |

ICD-9 = International Classification of Diseases, 9th Revision; ICD-10 = International Statistical Classification of Diseases and Related Health Problems, 10th Revision.

## 9.3.2.3 Review of patient profiles and medical records

The prescribed indication for olodaterol and indacaterol and the potential for off-label prescribing of these medications will be further evaluated through the clinical review of patient profiles of a random sample of about 100 new users of each medication prior to the first exposure to the respective drug. Patient profiles are chronological listings of the codes that represent clinical events recorded in the study databases for individual patients. These listings include general practitioner diagnoses, outpatient and hospital discharge diagnoses and procedures; and dispensings of medications. The clinical review of patient profiles will provide the most accurate information for evaluation of the indication and potential off-label use of olodaterol and indacaterol. This information will be useful for developing clinical algorithms that can be applied to the evaluation of all new users of olodaterol and indacaterol whose information is linked to general practitioner diagnoses.

The random sampling of patient profiles for review will be stratified by age (0-17 years, 18-39 years,  $\geq$  40 years) and sex because PPVs are expected to vary by prevalence of COPD, which in turn varies by age and sex.

#### 9.3.2.4 Classification of patients

According to the presence of a recorded diagnosis of COPD and/or asthma, new users of olodaterol and new users of indacaterol will be classified into the following categories: (1) on-label prescribing (indication of COPD), (2) off-label prescribing for asthma, and (3) off-label prescribing with no evidence of COPD or asthma (Table 5).

The following fifth-digit subclassification is for use with category 493.0-493.2, 493.9: 0, unspecified; 1, with status asthmaticus; 2, with (acute) exacerbation

Proprietary confidential information © 2014 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Table 5 Classification of patients according to indication or off-label prescribing of olodaterol and indacaterol

| Recorded diagnosis <sup>1</sup> | On-Label<br>Prescribing:<br>Indication of<br>COPD | Off-Label<br>Prescribing for<br>Asthma | Potential Off-<br>Label Prescribing<br>Other than<br>Asthma |
|---|---|---|---|
| COPD | Yes | | |
| COPD and asthma | Yes | | |
| Asthma | | Yes | |
| No COPD, no asthma | | | Yes |

COPD = Chronic Obstructive Pulmonary Disease.

#### 9.3.3 Characterisation of new users of olodaterol and indacaterol

New users of olodaterol and new users of indacaterol will be characterised at the index date according to demographic variables, available data on lifestyle habits, comorbidity, and use of medications. Comorbidity will be ascertained through diagnosis codes and procedures recorded at any time before the index date. Use of medications will be ascertained for the 12 months before the index date.

In the following sections, we list the variables that will be used to characterise new users of olodaterol and new users of indacaterol. The variables will be assessed according to the availability of information in each study database (see Table 8 on page 30 for availability of variables of interest). Some of the variables (e.g., lifestyle habits or socioeconomic indicators) may be partially or completely unavailable in the study databases. We provide ICD-10 and ICD-9 codes for diagnoses and procedures and ATC codes for medications.

#### 9.3.3.1 Demographics and lifestyle habits at the index date

- Age
- Sex
- Calendar year
- Body mass index
- Smoking status
- Alcohol consumption
- Socioeconomic indicators or proxies (e.g., deprivation index, education level, postal code)

#### 9.3.3.2 Respiratory comorbidity and allergies

• Time since first diagnosis of COPD

Diagnosis recorded at any time before the index date or at the index date.

Proprietary confidential information © 2014 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

• Respiratory conditions recorded at any time before the index date (Table 6).

Time between the first recorded diagnosis of COPD in the database and the index date will be ascertained for new users of olodaterol and indacaterol.

Table 6 Respiratory comorbidity and allergies

| <b>Disease Description</b> | ICD-10 | ICD-9 |
|----------------------------|----------|---------------|
| COPD | J41-J44 | 491, 492, 496 |
| Chronic bronchitis | J41-J42 | 491 |
| Emphysema | J43 | 492 |
| Other COPD | J44 | 496 |
| Asthma | J45, J46 | 493 |
| Pneumonia | J09-J18 | 480-486 |
| Allergic rhinitis | J30 | 477 |

COPD = Chronic Obstructive Pulmonary Disease; ICD-10 = International Statistical Classification of Diseases and Related Health Problems, 10th Revision. ICD-9 = International Classification of Diseases, 9th Revision.

### 9.3.3.3 Severity of COPD

The guidelines of the Global Initiative for Chronic Obstructive Lung Disease (GOLD) recommend that physicians evaluate the severity of COPD and its impact on the health of patients by the combination of (1) the current level of symptoms, (2) the severity of the spirometric abnormality, and (3) the risk of exacerbations. [P13-02399] The presence of comorbidities also determines the severity of COPD and is a predictor of morbidity and mortality. According to these parameters, severity of COPD is classified in four severity groups as illustrated in Figure 2.

Proprietary confidential information © 2014 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Risk 4 C D ≥ 2 GOLD classification of 3 airflow limitation 2 Α В ≤ 1 1 mMRC 0-1 mMRC ≥ 2 **CAT < 10 CAT ≥ 10** 

# Exacerbation history

Risk

#### **COPD Severity Categories**

| Severity<br>Category | Characteristics | Spirometric<br>Classification | Exacerbations per Year | mMRC | CAT |
|---|---|---|---|---|---|
| A | Low risk, fewer symptoms | GOLD 1-2<br>(mild- | ≤ 1 | 0-1 | < 10 |
| В | Low risk, more symptoms | moderate) | | ≥ 2 | ≥ 10 |
| С | High risk, fewer symptoms | GOLD 3-4<br>(severe-very | ≥ 2 | 0-1 | < 10 |
| D | High risk, more symptoms | severe | | ≥ 2 | ≥ 10 |

CAT = COPD Assessment Test; COPD = Chronic Obstructive Pulmonary Disease; GOLD = Global Initiative for Chronic Obstructive Lung Disease; mMRC = Modified British Medical Research Council Questionnaire.

Source: Adapted from GOLD, 2013. [P13-02399]

Figure 2 Association between symptoms, spirometric classification, and future risk of exacerbations according to the Global Initiative for Obstructive Lung Disease

Some of the parameters to evaluate the severity of COPD are not available or are only partially recorded in automated health databases. These parameters include the level of symptoms of COPD and the results from spirometric tests. Therefore, severity of COPD in studies conducted in health databases is usually evaluated by other parameters that serve as proxies of severity. [R08-1492] [R09-0579] [R13-1392] [P09-04948] [P11-13226]

A summary of the evaluation of severity of COPD in health database studies is presented in ANNEX 3. In a study conducted in the General Practice Research Database (now known as the Current Practice Research Database) from the United Kingdom, the definition of severity was based on the intensity of use of bronchodilators and the use of oxygen therapy or nebulised therapy.[R08-1492] A modification of this definition of severity was used in a recent study conducted in the Integrated Primary Care Information Project database in the Netherlands.[P11-13226] The definition used in that study included hospitalisations for COPD, the use of antibiotics for the treatment of respiratory tract infections, and the use of systemic glucocorticosteroids for the treatment of COPD exacerbations. The classification of severity based on these factors had a PPV of 82% when compared with results from spirometry. In another study conducted in the Saskatchewan Health databases in Canada, determinants of COPD severity were the presence of emphysema, the use of nebuliser therapy, the use of oxygen therapy, the use of inhaled and/or systemic glucocorticosteroids, the intensity of bronchodilator use, pneumonia, and prior COPD exacerbation.[R09-0579] These factors were associated with increased cardiovascular morbidity and mortality.

**BI Study Number 1222.53** 

Proprietary confidential information © 2014 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## 9.3.3.4 Definition of COPD severity

Severity of COPD will be evaluated among new users of olodaterol and indacaterol that have a recorded diagnosis of COPD before the index date. Severity of COPD will be evaluated at the index date by a modified version of the algorithm developed by Verhamme and colleagues [P11-13226] (see Table 7).

Table 7 Definition criteria of COPD severity

| Severity of COPD | Definition |
|---|---|
| Mild | Less than 2 dispensings of the same COPD drug class with a maximum interval of 6 months in the 12 months before the index date. |
| Moderate | Regular bronchodilator treatment, defined as having at least 2 dispensings of the same COPD drug class with a maximum interval of 6 months in the 12 months before the index date <sup>1,2</sup> |
| Severe | Occurrence of at least one of the following events in the year before the index date: |
| | • Hospitalisation for COPD <sup>2</sup> |
| | <ul> <li>Recorded diagnosis of pneumonia<sup>2</sup></li> </ul> |
| | • Third course of antibiotics for respiratory tract infections <sup>2</sup> |
| | • Second course of systemic corticosteroids for the treatment of COPD exacerbation <sup>2</sup> |
| Very severe | Occurrence of at least one of the following events in the year before the index date unless other time period is specified: |
| | • Dispensed oxygen therapy <sup>1,2</sup> |
| | • Dispensed nebuliser therapy <sup>1,2</sup> |
| | • Diagnosis of emphysema at any time before the index date <sup>2</sup> |

COPD = Chronic Obstructive Pulmonary Disease.

Sources: modified from Verhamme et al., 2012 [P11-13226]; Soriano et al., 2001 [R08-1492]; and Curkendall et al., 2006. [P07-09136]

- 1 Severity criteria also included in definition from Soriano et al., 2001. [R08-1492]
- 2 Severity criteria also included in definition from Curkendall et al., 2006. [P07-09136]

The use of antibiotics and oral corticosteroids and hospitalisations for COPD haven been used by other authors as markers of severity of COPD exacerbations. [P12-09396] [P12-09395] [P12-14293]

The operational definitions to be applied when assessing the severity of COPD are as follows:

- Same-class bronchodilators. The following bronchodilators classes will be considered (see Annex Table 4:2):
  - Inhaled short-acting muscarinic antagonists (SAMAs)
  - Inhaled long-acting muscarinic antagonists (LAMAs)

I Study Number 1222.53 c02329987-02

Proprietary confidential information © 2014 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

- Inhaled short-acting beta2-agonists (SABAs)
- Inhaled LABAs
- Inhaled glucocorticosteroids (ICSs)
- Fixed combinations of SABAs and SAMAs
- Fixed combinations of SABAs and ICSs
- Fixed combinations of LABAs and ICSs
- Systemic glucocorticosteroids
- Systemic beta2-agonists
- Xanthines
- Roflumilast
- Hospitalisation for COPD
  - Primary or secondary hospital discharge diagnosis for COPD
  - ICD-10 codes: J40-J44; ICD-9 codes: 491, 492, 496
- Recorded diagnosis of pneumonia
  - Primary or secondary hospital discharge diagnosis for pneumonia
  - ICD-10 codes J09-J18; ICD-9 codes: 480-486
- Third course of antibiotics for respiratory tract infections
  - A course with antibiotic is defined as that involving consecutive dispensings of antibiotics with less than 7 days between the end of days of supply of one dispensing and the date of the next dispensing
  - ATC codes for antibiotics: J01 (antibacterials for systemic use)
- Second course of systemic glucocorticosteroids for the treatment of COPD exacerbation
  - A course with systemic corticosteroids is defined as that involving consecutive dispensings with less than 7 days between the end of days of supply of one dispensing and the date of the next dispensing.
  - ATC codes for systemic glucocorticosteroids: H02AB
- Oxygen therapy, ATC code: V03AN01
- Nebuliser therapy (to be identified in each database using national drug codes)
- Primary or secondary hospital outpatient or inpatient discharge diagnosis of emphysema at any time before the index date
  - ICD-10 code: J43; ICD-9 code: 492

## 9.3.3.5 Other comorbidity and conditions

The following comorbidities and conditions recorded at any time before the index date will be evaluated: cardiovascular diseases, hyperlipidaemia, diabetes mellitus, renal disease,

Proprietary confidential information © 2014 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

anaemias, peptic ulcer disease, liver disease, osteoporosis, rheumatoid arthritis, systemic connective tissue diseases, malignancy, depressive disorders, and pregnancy. Specific diseases and conditions and ICD-10 and ICD-9 codes are provided in Annex 4, Annex Table 4:1

#### 9.3.3.6 Comedications

The following comedications dispensed within 12 months before the index date will be evaluated: respiratory medications, cardiovascular medications, antithrombotic agents, systemic antibacterials, iron preparations, proton pump inhibitors, drugs used in diabetes, drugs for musculoskeletal system conditions, antidepressants, antineoplastic agents, immunosuppressants, antivirals for systemic use, hormone-replacement therapy, and drugs used in nicotine dependence.

Specific medications and ATC codes are provided in Annex Table 4:2.

#### 9.3.3.7 Health care resource utilisation

Health care resource utilisation will be evaluated for the **12 months before the index date**.

- Total number of dispensing; all medications included in Annex Table 4:2
- Total number of dispensings for respiratory medications; all medications included in the section of respiratory medications in Annex Table 4:2
- Total number of dispensings for systemic glucocorticosteroids; ATC code H02AB
- Total number of dispensings for LABAs; ATC codes R03AC012 (salmeterol) and R03AC013 (formoterol)
- Total number of hospitalisations; number of hospitalisations for any cause
- Total number of hospitalisations for COPD; number of hospitalisations with a primary discharge code for COPD; ICD-10 codes J40-J44; ICD-9 codes: 491, 492, 496
- Total number of hospitalisations for asthma; number hospitalisations with a primary discharge code for asthma; ICD-10 codes J45, J46; ICD-9 code: 493

## 9.3.4 Outcomes

### 9.3.4.1 Primary outcome

The primary outcome is the prevalence of off-label prescribing among new users of olodaterol.

Proprietary confidential information © 2014 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 9.3.4.2 Secondary outcomes

9.3.4.3 The secondary outcome is the prevalence of off-label prescribing among new users of indacaterol

#### 9.3.5 Covariates

Not applicable.

#### 9.4 DATA SOURCES

The study will be conducted in the following databases:

- PHARMO Database Network
- National Registers in Denmark
- National Registers in Sweden

A description of each database is provided in the following sections; further details are provided from the feasibility report, dated 1 November 2013, and in ANNEX 5. The study will be conducted by using data on drug dispensings and disease occurrence routinely collected on an ongoing basis for large population-based automated health care databases in the Netherlands, Denmark, and Sweden (see Table 1 and Table 2 for characteristics of these databases). New users will be characterised in terms of past medical history and use of medications. Off-label prescribing will be evaluated for those new users for whom general practitioner diagnoses are available. An overview of the information on diagnoses and procedures by data source is shown in the table below (Table 8).

#### 9.4.1 PHARMO Database Network

#### 9.4.1.1 Database characteristics

The PHARMO Database Network consists of multiple databases containing data files on approximately 3.2 million community-dwelling inhabitants in geographically defined areas covering approximately 20% of the Netherlands. Data sources include information from general practitioners (GPs), community pharmacies, hospitals, and laboratory sources.

The patients covered in each database are not necessarily included in all of the databases, as some of the geographical areas overlap partially, but if they are in more than one database, they can be linked to construct the medical history as shown in Figure 3. Thus, high-quality research can be conducted with ascertainment of patient demographics, drug dispensings, hospital morbidity, clinical laboratory results, and date of death.

The dispensing (outpatient pharmacy) database covering 3.2 million individuals can use a validated algorithm to identify patients with COPD, asthma, or other respiratory conditions. All patients are linked with the hospitalisation database (100% overlap between outpatient

Proprietary confidential information © 2014 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

and hospitalisation database). Approximately 440,000 patients can be linked to GP data for severity indicators as recorded by the GP.



Figure 3 Schematic overview of overlap example among databases included in the PHARMO Database Network

The GP database covering 1.4 million individuals has information as recorded by the GP, including forced expiratory volume in 1 second (FEV<sub>1</sub>) and spirometry data. Approximately half of the population (440,000) in the GP database can be linked to both dispensing (outpatient pharmacy) and hospitalisation data.

#### 9.4.2 Denmark

The Danish health care system provides universal coverage to all Danish residents (5.5 million inhabitants). Health care coverage includes visits to GPs and specialists, hospital admissions, and outpatient visits. The costs of medicines are partially covered by the Danish health system. The centralised Civil Registration System in Denmark allows for personal identification of each person in the entire Danish population and for the possibility of linkage to all Danish registries containing civil registration numbers, such as the Danish National Registry of Patients, Danish National Prescription Database, the Prescription Databases of the Central Denmark Region, and the Danish Registry of Causes of Death. Data collected in these registries are available for research purposes. The availability of the Danish General Practice Database (DAMD) is a recent development in the group of Danish databases used for research. It provides information from selected general practices nationwide, with the purposes of promoting and improving the quality of care in general practice and providing data for research concerning general practice. [R13-5415] The DAMD currently covers about 1 million population.

For 1980-2008, The National Registry of Patients counted 236,494 patients with a first hospital contact for COPD. [R12-3324] From the National Health Service, for persons aged 45 to 84 years, the prevalence of COPD was estimated at 12%, using a sample of 299,000 residents of two counties. [R12-3265]

#### 9.4.3 Sweden

Since 1987, Sweden has mandated collection of hospital care data nationally; same-day surgery and psychiatric care have since been added to the database. [R14-0444] The hospital data are held in the Swedish National Patient Register (NPR) (sometimes called the Hospital Discharge Register), along with a Cause of Death Register. The Swedish NPR comprises all admissions to hospital care and hospital outpatient diagnoses. Primary and several secondary

Proprietary confidential information © 2014 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

diagnoses are recorded. With the national personal identification number, patients can be tracked over time and from one hospital to another. As of 2004, few admissions were missing a personal identification number; for example, for stroke, 0.5% of hospitalisations lacked an identification number in a study of two counties. For acute hospital care, more than 99% of the hospital stays had at least a primary diagnosis recorded. [R14-0356] A validation review of the NPR by the National Board of Health and Welfare showed that 85% to 95% of all diagnoses are valid. [R14-0357]

Primary care data in Sweden may be available for the counties of Stockholm and Göteborg through the County Council health registers. The population of these two counties covers approximately 25% of the total Swedish population.

Ascertained from the Obstructive Lung Disease in Northern Sweden study, the prevalence of patients with diagnosed COPD in a subset of the study cohort and aged 46 years or older was 14.3%, when evaluated by GOLD criteria, and 8.1% when evaluated by British Thoracic Society criteria. [R13-1576] From the National Oxygen Register, the estimated number of patients with severe COPD was 8,712. [R14-0353]

### 9.4.4 Summary of study databases

Table 8 shows and compares the characteristics of the study databases.

Table 8 Overview of the study databases

| Data Element | PHARMO<br>(Netherlands) | National Registers,<br>Denmark | National Registers,<br>Sweden |
|---|---|---|---|
| Database type | Patient-centric data obtained from community pharmacies and with variable linkage rates to other health care files | National health record and prescription databases linked through the unique civil personal registration number | National health<br>record databases<br>capable of linkage<br>through the unique<br>civil personal<br>registration number |
| Database population | 3.2 million | Denmark | Sweden |
| Country population <sup>1</sup> | 16,779,575 | 5,602,628 | 9,555,893 |
| Approximate proportion of the country's population covered by the database | 20% | 100% | 100% |

Proprietary confidential information © 2014 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Table 8 (con't) Overview of the study databases

| Data Element | PHARMO<br>(Netherlands) | National Registers,<br>Denmark | National Registers,<br>Sweden |
|---|---|---|---|
| Representative-<br>ness of patients<br>and practices | Known to be representative [ <u>P93-73309</u> ] [ <u>P14-01899</u> ] | Complete, given that<br>the total country<br>population is<br>included | Complete, given that<br>the total country<br>population is<br>included |
| Data on medications | Dispensings from community pharmacies and prescriptions from GP database | Pharmacy-dispensed prescriptions | All pharmacy-<br>dispensed<br>prescriptions |
| Dose | Yes | Formulation strength | Formulation strength |
| Duration | Yes | Based on prescriptions | Based on dispensed prescriptions |
| Drug dictionary codes/therapeutic classification | ATC | ATC | ATC |
| Indacaterol | 4,000 | 47,400 (2010-2011) | 6,361 (2010-2011) |
| Number of users of indacaterol | 1,200 | 6,093 (2010-2011) | 110 (2010)<br>2,565 (2011) |
| Clinical indication | For approximately 440,000 PHARMO subjects (included in outpatient database), via linkage to GP files and proximity of clinical diagnoses; for all subjects in GP database | Not recorded but may<br>be surmised based on<br>GP diagnoses for GP-<br>linked practices and<br>proxies (i.e.,<br>prescribed<br>medication and<br>hospital discharge<br>diagnosis history) for<br>not-linked practices | Not recorded but<br>may be surmised<br>based on GP<br>diagnoses for GP-<br>linked practices and<br>proxies (i.e.,<br>prescribed<br>medication and<br>hospital discharge<br>diagnosis history) for<br>not-linked practices |
| Prescriber characteristics | GP vs. specialist | GP vs. specialist | Profession Level of education Speciality |

Proprietary confidential information © 2014 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Table 8 (con't) Overview of the study databases

| Data Element | PHARMO<br>(Netherlands) | National Registers,<br>Denmark | National Registers,<br>Sweden |
|---|---|---|---|
| Outpatient diagnosis | For all PHARMO subjects (included in outpatient databases): main diagnoses in ICD-9-CM for all admissions for > 24 hours and admissions for < 24 hours for which a bed is required; for subcohort of GP database patients with linkage to outpatient pharmacy database | Hospital outpatient diagnoses General practitioner diagnoses for about 1 million population recorded via ICPC coding | Hospital diagnoses. General practitioner diagnoses for the counties for Stockholm and Göteborg recorded via ICPC coding |
| Hospital<br>diagnosis | Main hospital diagnostic/surgical procedures | Yes | Yes |
| Procedure codes | Available for approximately 1 million of pharmacy file patients; GP laboratory tests for all patients in GP database | Yes, ICD-10 | Yes, NCSP version<br>1.16:2012 |
| Pulmonary<br>function testing | With difficulty | From hospital clinics<br>and also from<br>primary care when<br>recorded | From hospital clinics<br>and also from<br>primary care when<br>recorded |
| Information on death | Fact and date of death, Mortality Register | Fact, date, and<br>underlying cause of<br>death available in<br>National Death<br>Register | Fact, date, and<br>underlying cause of<br>death available in<br>National Death<br>Register |
| Access to medical records | Variable | No | No |

Proprietary confidential information © 2014 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Table 8 (con't) Overview of the study databases

| Data Element | PHARMO<br>(Netherlands) | National Registers,<br>Denmark | National Registers,<br>Sweden |
|---|---|---|---|
| Lifestyle risk<br>factors (smoking<br>status, BMI,<br>alcohol intake) | Yes, if recorded by GPs | Yes, if recorded by GPs | Yes, if recorded by GPs |
| Data availability | Annual | Since 1994 | Since 2005 |
| Updates | Pharmacy data: 2<br>months<br>All other data:<br>annual; available<br>following Q3-Q4 | Annual | Annual |
| Approximate time lag | No | 1 year | 2012 data will be<br>available in 3Q-4Q<br>2013 |
| Data transfer | Review by the independent compliance committee STIZON/PHARMO Institute This committee consists of representatives of the individual data suppliers and is chaired by a privacy expert | No, requires collaboration with local investigator | No, requires collaboration with local investigator |
| Approval process | Data application and ethics committee approval required | Data application and ethics committee approval required | Data application and ethics committee approval required |

ATC = Anatomical Therapeutic Chemical; BMI = Body Mass Index; GP = General Practitioner; ICD-9-CM = International Classification of Diseases, 9th Revision, Clinical Modification; ICD-10 = International Statistical Classification of Diseases and Related Health Problems, 10th Revision; ICD-10-CM = International Classification of Diseases, 10th Revision, Clinical Modification; ICPC = International Classification of Primary Care; NCSP = Nordic Medico-Statistical Committee's Classification of Surgical Procedures.

## 9.5 STUDY SIZE

Actual counts of numbers of patients using olodaterol in European countries are not yet available. Table 9 shows the confidence intervals around estimated prevalence of comorbidity and comedications under various exposure group size scenarios.

Eurostat. 2013. Available at: website: epp.eurostat.ec.europa.eu/tgm/table.do?tab=table&init=1&language=en&pcode=tps00001&plugin=1. Accessed January 28, 2014.

Proprietary confidential information © 2014 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Table 9 Confidence intervals around selected estimated prevalences for varying numbers of patients

| Number of | 95% Confidence Intervals for Various Prevalences of Diseases (%) | | | | |
|---|---|---|---|---|---|
| Patients | 1% | 2% | 5% | 7% | 10% |
| 300 | 0.2-2.9 | 0.7-4.3 | 2.8-8.1 | 4.4-10.5 | 6.8-14.0 |
| 800 | 0.4-2.0 | 1.1-3.2 | 3.6-6.7 | 5.3-9.0 | 8.0-12.3 |
| 2,000 | 0.6-1.5 | 1.4-2.7 | 4.1-6.0 | 5.9-8.2 | 8.7-11.4 |
| 5,000 | 0.7-1.3 | 1.6-2.4 | 4.4-5.6 | 6.3-7.7 | 9.2-10.9 |

Note: This table was prepared with the use of Episheet—spreadsheets for the analysis of epidemiologic data. [R13-1396]

A small number of users of olodaterol in each database during the first years (2014-2016) after launch may result in imprecise prevalence estimates for conditions with a prevalence of 10% and below, especially when stratified analyses are conducted.

#### 9.6 DATA MANAGEMENT

Routine procedures include checking electronic files, maintaining security and data confidentiality, following analysis plans, and performing quality-control checks of all programs. Each database research partner will maintain any patient-identifying information securely onsite according to internal standard operating procedures.

Each collaborating data source has been reviewed and qualified by the RTI Health Solutions Office of Quality Assurance. Each research team will follow its own established procedures and generate appropriate result tables. All summary tables of results, and no individual patient identifiers, will be provided to RTI Health Solutions, which will compile the results and develop the report. RTI Health Solutions will follow quality-control procedures regarding transfer of data.

Security processes will be in place to ensure the safety of all systems and data. Every effort will be made to ensure that data are kept secure so that they cannot be accessed by anyone except select study staff.

Appropriate data storage and archiving procedures will be followed. Standard procedures will be in place at each location handling the data to restore files in the event of a hardware or software failure.

The extent of missing data will be evaluated and described. Due to the nature of this study, no imputation of missing data is planned.

For requests to access to data for audit purposes, only aggregated data from all research centres will be available at the coordinating centre. The audit trail will consist of a detailed description of the methods to extract and process the electronic health records or claims data, as applicable. Access to raw data at each database research centre will require the data

Proprietary confidential information © 2014 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

requestor to obtain a license or apply for approval at a research committee and to fulfil the conditions required under the governance rules of each database research centre.

#### 9.7 DATA ANALYSIS

All analyses will be conducted separately in each study database and will be further analysed separately by new users of olodaterol and by new users of indacaterol, further stratified by treatment-naïve subjects and switchers. Analyses will be conducted annually for three consecutive years. Each year will include all patients starting treatment with olodaterol or indacaterol in that specific year. Statistical analyses will be descriptive in nature. Descriptive statistics will include the absolute and relative number of subjects, mean, median, standard deviation, and range for continuous variables. Statistical inference will not be performed (e.g., no *P* values will be generated).

## 9.7.1 Main analysis

# 9.7.2 Indication and potential off-label prescribing

Number and proportion of new users for each indication (COPD only, COPD and asthma, asthma only, and no COPD or asthma) associated with the initiation of treatment.

This analysis will be conducted using data linked to diagnoses recorded by general practitioners (primary care information):

- PHARMO-GP, covering about 440,000 population
- Danish General Practice Database, covering about 1 million population
- Swedish General Practice Database for the counties of Stockholm and Göteborg

#### 9.7.3 Number of users and patterns of use

The following analyses will be conducted:

**Dose at the start date**: Dose at the start date will be ascertained by the dispensed DDD and the estimation of the daily dose. The estimated daily dose dispensed at the index date will be calculated using the recorded information on strength and quantity dispensed and the days of supply of the first prescription for olodaterol and indacaterol. The mean (SD) number of packages and daily dose will be calculated.

**Age and sex distribution of users at the index date**: Number and percentage of users of olodaterol and indacaterol at the index date by sex and the following groups of age (in years): 0-17, 18 to 29, 30 to 39, 40 to 49, 50 to 59, 60 to 69, 70 to 79, 80 or older.

#### 9.7.4 Characterisation of new users at the index date

The number and percentage of each variable of interest (as specified in Section 9.3) at the index date will be estimated separately among new users of olodaterol and among new users of indacaterol. All analyses will be stratified by the following variables:

• Age in years, categorised as 0 to 17 years, 18 to 39 years, and 40 years or older
Proprietary confidential information © 2014 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

- Sex
- Switchers at the index date (as defined in Section 9.2.3) and treatment-naïve subjects
- Indication
  - COPD only
  - COPD and asthma
  - Asthma only
  - Neither COPD nor asthma
- Calendar year of index date: 2014, 2015, 2016

The following analyses will be performed:

**Time since first recorded diagnosis of COPD**: Mean (SD), median, 25th percentile, and 75th percentile.

**Lifestyle habits**: Distribution of new users by categories of body mass index, smoking status, alcohol consumption, and socioeconomic status at the index date, according to the type of information available in each database.

**Respiratory comorbidity and allergies**: Number and proportion of new users with at least one diagnosis for each respiratory condition listed in Table 5 that was recorded at any time before the index date.

**Severity of COPD**: Number and proportion of new users for each category of severity of COPD: mild, moderate, severe, and very severe.

**Other comorbidity**: Number and proportion of patients with at least one diagnosis for each of the comorbidity conditions listed in Table 8 and recorded at any time before the index date.

**Comedications**. Number and proportion of patients with at least one dispensing for each of the medications listed in Annex Table 4:2 taking place in the 12 months before the index date.

**Health care resources utilisation**: Distribution of new users as defined by the following categories of variables evaluated within the 12 months before the index date:

- Total number of dispensings: 0, 1 to 4, 5 to 9, 10 or more
- Total number of dispensings for respiratory medications (Annex Table 4:2): 0, 1 to 4, 5 to 9, 10 or more
- Total number of dispensings for systemic glucocorticosteroids: 0, 1 to 4, 5 to 9, 10 or more
- Total number of dispensings for LABAs: 0, 1 to 4, 5 to 9, 10 or more
- Total number of hospitalisations: 0, 1, 2, 3 to 4, 5 or more
- Total number of hospitalisations for COPD: 0, 1, 2, 3 to 4, 5 or more
- Total number of hospitalisations for asthma: 0, 1, 2, 3 to 4, 5 or more

Proprietary confidential information © 2014 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 9.8 QUALITY CONTROL

At the coordinating centre, an independent Office of Quality Assurance performs audits and assessments that involve various aspects of its projects, including but not limited to documentation of education and training, data entry, data transfer, and approval of the institutional review board at RTI International, of which RTI Health Solutions is a research unit. Such audits at RTI Health Solutions will be conducted by the Office of Quality Assurance according to established criteria in standard operating procedures and other applicable procedures. Each of the database research centres will follow its own quality and audit trail procedures. The quality and audit trails at each centre may be different.

Data management and analysis will be conducted in each database. Standard operating procedures at each database will be used to guide the conduct of the study. These procedures include internal quality audits and the opportunity for external audits, rules for secure and confidential data storage, methods to maintain and archive project documents, quality-control procedures for programming, standards for writing analysis plans, and requirements for senior scientific review. RTI Health Solutions will follow quality-control procedures for report generation, including senior review by an expert other than the author.

#### 9.9 LIMITATIONS OF THE RESEARCH METHODS

Existing population-based data are very useful for evaluating research questions about real-world clinical practice because of the diversity of patients and medical practices represented therein. However, the results must be interpreted with caution because such data sources are known to misclassify information of interest, in the following ways:

- The length of medical history in some databases will be limited, and earlier medical events or drug exposures may be unknown. Therefore, the prevalence of some conditions may be underestimated.
- Information on prescriber characteristics is likely to be limited in some of the available databases.
- Clinical differential diagnosis between COPD and asthma might be difficult, and it is even more challenging to differentiate these conditions in database studies.
- For severity of COPD, ideally FEV<sub>1</sub> would be useful to classify all individuals by application of standard criteria; however, it is anticipated that this information is not recorded systematically in the study databases. Therefore, classification of severity of COPD in database studies uses proxies, such as use of COPD medications and use of health care services.
- For Denmark and Sweden, this study will be conducted by researchers affiliated with institutions that have access to the national registers. Thus, the conduct of the study in these countries will depend on the scientific and regulatory interest of these researchers, as well as on their availability during the study period.
- Study size depends upon the uptake of olodaterol.

Proprietary confidential information © 2014 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 9.10 OTHER ASPECTS

#### 9.10.1 Bias

The use of hospital outpatient and/or inpatient discharge diagnoses can overestimate potential off-label prescribing. For this reason, and because use of hospital discharge diagnoses does not ascertain patients diagnosed with COPD who are not hospitalised, off-label use will be assessed in the subset of new users linked to the general practice (primary care) registers. In the three countries primary care data are only available for a subset of the population.

Proprietary confidential information © 2014 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 10. PROTECTION OF HUMAN SUBJECTS

The study will be conducted in accordance with the International Society for Pharmacoepidemiology's *Guidelines for Good Pharmacoepidemiology Practices* [R11-4318] and in accordance with the European Network of Centres for Pharmacoepidemiology and Pharmacoepidemiology. [R13-5419] The ENCePP *Checklist for Study Protocols* [R13-1395] is completed (see ANNEX 2), and the study will be registered in the EU PAS Register. [R14-0354]

The study is a drug utilisation study and will comply with the definition of the non-interventional (observational) study provided in the 2012 *Guideline on Good Pharmacovigilance Practice: Module VIII—Post-Authorisation Safety Studies.* [R13-5420]. The study will comply with the nature of non-interventional (observational) studies referred to in the International Conference on Harmonisation's harmonised tripartite guideline *Pharmacovigilance Planning E2E.* [R11-2259]

Proprietary confidential information © 2014 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## 11. MANAGEMENT AND REPORTING OF ADVERSE EVENTS/ADVERSE REACTIONS

Based on current guidelines from the International Society for Pharmacoepidemiology [R11-4318] and the European Medicines Agency (EMA) *Guideline on Good Pharmacovigilance Practices (GVP) Module VI - Management and Reporting of Adverse Reactions to Medicinal Products*, [R13-1970] non-interventional studies such as the one described in this protocol conducted using aggregated patient data from electronic health care records do not require expedited reporting of suspected adverse events/reactions. Based on the data planned for this study, no suspected adverse events/reactions are expected.

Proprietary confidential information © 2014 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## 12. PLANS FOR DISSEMINATING AND COMMUNICATING STUDY RESULTS

The study protocol synopsis, study status, and report(s) will be included in regulatory communications in line with the risk management plan, Benefit-Risk Evaluation Report, and other regulatory milestones and requirements.

Study results will be published following the International Committee of Medical Journal Editors recommendations, [R13-5418] and communication in appropriate scientific venues (e.g., the International Society for Pharmacoepidemiology) will be considered.

When reporting results of this study, the appropriate Strengthening the Reporting of Observational Studies in Epidemiology checklist [R11-4902] will be followed.

### 13. REFERENCES

### 13.1 PUBLISHED REFERENCES

| P07-09136 | Curkendall SM, Lanes S, de Luise C, Stang MR, Jones JK, She D, et al. Chronic obstructive pulmonary disease severity and cardiovascular outcomes. Eur J Epidemiol. 2006;21(11):803-13. |
|---|---|
| P09-04948 | Ogale SS, Lee TA, Au DH, Boudreau DM, Sullivan SD. Cardiovascular events associated with ipratropium bromide in COPD. Chest. 2010 Jan;137(1):13-9. |
| P11-13226 | Verhamme KM, Afonso AS, van Noord C, Haag MD, Koudstaal PJ, Brusselle GG, et al. Tiotropium Handihaler and the risk of cardio- or cerebrovascular events and mortality in patients with COPD. Pulm Pharmacol Ther. 2012 Feb;25(1):19-26. |
| P12-09395 | Wilchesky M, Ernst P, Brophy JM, Platt RW, Suissa S. Bronchodilator use and the risk of arrhythmia in COPD: part 1: Saskatchewan cohort study. Chest. 2012 Aug;142(2):298-304. |
| P12-09396 | Wilchesky M, Ernst P, Brophy JM, Platt RW, Suissa S. Bronchodilator use and the risk of arrhythmia in COPD: part 2: reassessment in the larger Quebec cohort. Chest. 2012 Aug;142(2):305-11. |
| P12-14293 | Suissa S, Dell'Aniello S, Ernst P. Long-term natural history of chronic obstructive pulmonary disease: severe exacerbations and mortality. Thorax. 2012 Nov;67(11):957-63. |
| P13-02399 | GOLD. Global strategy for the diagnosis, management, and prevention of chronic obstructive pulmonary disease. Updated 2013. Global Initiative for Chronic Obstructive Lung Disease; 2013. Available at: website: goldcopd.org/guidelines-global-strategy-for-diagnosis-management.html. Accessed 17 October 2013. |
| P14-01899 | Herings RMC, Pedersen L. Pharmacy-based medical record linkage systems. In: Strom BL KS, Hennessy S, editor. Pharmacoepidemiology, 5th edition. 5th ed: John Wiley & Sons, Ltd.; 2012. p. 270-86. |
| P93-73309 | Herings RM, Bakker A, Stricker BH, Nap G. Pharmaco-morbidity linkage: a feasibility study comparing morbidity in two pharmacy based exposure cohorts. J Epidemiol Community Health. 1992 Apr;46(2):136-40. |

**BI Study Number 1222.53** 

R12-3324

Proprietary confidential information © 2014 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

R06-4117 Halbert RJ, Natoli JL, Gano A, Badamgarav E, Buist AS, Mannino DM. Global burden of COPD: systematic review and metaanalysis. Eur Respir J. 2006 Sep;28(3):523-32. Soriano JB, Visick GT, Muellerova H, Payvandi N, Hansell AL. R07-2620 Patterns of comorbidities in newly diagnosed COPD and asthma in primary care. Chest. 2005 Oct;128(4):2099-107. R08-1492 Soriano JB, Maier WC, Visick G, Pride NB. Validation of general practitioner-diagnosed COPD in the UK General Practice Research Database. Eur J Epidemiol. 2001;17(12):1075-80. Curkendall SM, DeLuise C, Jones JK, Lanes S, Stang MR, R09-0579 Goehring E, Jr., et al. Cardiovascular disease in patients with chronic obstructive pulmonary disease. Saskatchewan Canada cardiovascular disease in COPD patients. Ann Epidemiol. 2006 Jan;16(1):63-70. WHO. The global burden of disease: 2004 update. Table 7. R09-2531 Geneva: World Health Organization, Department of Health Statistics and Informatics; 2008. Available at: website: who.int/healthinfo/global burden disease/GBD report 2004updat e full.pdf. Accessed 14 November 2013. R11-2259 ICH. Technical requirements for registration of pharmaceuticals for human use. Pharmacovigilance planning. E2E. International Conference on Harmonisation; November 2004 2004. Available at: website: ich.org/products/guidelines/efficacy/efficacysingle/article/pharmacovigilance-planning.html. Accessed 26 July 2012. ISPE. Guidelines for good pharmacoepidemiology practices (GPP). R11-4318 International Society for Pharmacoepidemiology; April 2007 2007. Available at: website: pharmacoepi.org/resources.guidelines 08027.cfm. Accessed 01 March 2013. R11-4902 STROBE. STROBE checklist. Strengthening the Reporting of Observational Studies in Epidemiology; 2007. Available at: website: strobe-statement.org/index.php?id=available-checklists. Accessed 01 March 2013. R12-3265 Hansen JG, Pedersen L, Overvad K, Omland O, Jensen HK, Sorensen HT. The Prevalence of chronic obstructive pulmonary disease among Danes aged 45-84 years: population-based study. COPD. 2008 Dec;5(6):347-52.

Kornum JB, Svaerke C, Thomsen RW, Lange P, Sorensen HT. Chronic obstructive pulmonary disease and cancer risk: a Danish

R13-5420

Proprietary confidential information © 2014 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

nationwide cohort study. Respir Med. 2012 Jun;106(6):845-52. Eisner MD, Omachi TA, Katz PP, Yelin EH, Iribarren C, Blanc R13-1392 PD. Measurement of COPD severity using a survey-based score: validation in a clinically and physiologically characterized cohort. Chest. 2010 Apr;137(4):846-51. ENCePP. ENCePP checklist for study protocols (revision 2). R13-1395 European Network of Centres for Pharmacoepidemiology and Pharmacovigilance; 14 January 2013. Available at: website: encepp.eu/standards and guidances/checkListProtocols.shtml. Accessed 8 January 2014. R13-1396 Rothman KJ. Episheet--spreadsheets for the analysis of epidemiologic data. October 25, 2011, version. 2011. Available at: website: epidemiolog.net/studymat/. Accessed 14 February 2013. Lindberg A, Bjerg A, Ronmark E, Larsson LG, Lundback B. R13-1576 Prevalence and underdiagnosis of COPD by disease severity and the attributable fraction of smoking Report from the Obstructive Lung Disease in Northern Sweden Studies. Respir Med. 2006 Feb;100(2):264-72. R13-1970 EMA. Guideline on good pharmacovigilance practices (GVP). Module VI – Management and reporting of adverse reactions to medicinal products. European Medicines Agency; 22 June 2012. Available at: website: emea.europa.eu/docs/en GB/document library/Scientific guidelin e/2012/06/WC500129135.pdf. Accessed 8 January 2014. R13-5415 Danish Quality Unit of General Practice. Danish General Practice Database (DAMD). 2014. Available at: website: dake.dk/flx/english/dak e it/danish general practice database damd/ . Accessed 31 January. R13-5418 ICMJE. Recommendations for the conduct, reporting, editing, and publication of scholarly work in medical journals. International Committee of Medical Journal Editors; August 2013. Available at: website: icmje.org/urm main.html. Accessed 28 October 2013. R13-5419 ENCePP. Guide on methodological standards in pharmacoepidemiology (revision 2). EMA/95098/2010 Rev.2. European Network of Centres for Pharmacoepidemiology and Pharmacovigilance; 18 June 2013. Available at: website: encepp.eu/standards and guidances/methodologicalGuide.shtml. Accessed 8 January 2014.

EMA. Guideline on good pharmacovigilance practices (GVP).

| 1 Toprictary confider | tital information © 2014 Bochinger ingenienti international Gillott of one of more of its armiated comp |
|---|---|
| | Module VIII – Post-authorisation safety studies (EMA/813938/2011 Rev 1). European Medicines Agency; 19 April 2013. Available at: website: emea.europa.eu/docs/en_GB/document_library/Scientific_guidelin e/2012/06/WC500129137.pdf. Accessed 8 January 2014. |
| R14-0349 | Örtqvist AK, Lundholm C, Wettermark B, Ludvigsson JF, Ye W, Almqvist C. Validation of asthma and eczema in population-based Swedish drug and patient registers. Pharmacoepidemiol Drug Saf. 2013 Aug;22(8):850-60. |
| R14-0350 | Marsh SE, Travers J, Weatherall M, Williams MV, Aldington S, Shirtcliffe PM, et al. Proportional classifications of COPD phenotypes. Thorax. 2008 Sep;63(9):761-7. |
| R14-0351 | Juhn Y, Kung A, Voigt R, Johnson S. Characterisation of children's asthma status by ICD-9 code and criteria-based medical record review. Prim Care Respir J. 2011 Mar;20(1):79-83. |
| R14-0352 | Blais L, Lemiere C, Menzies D, Berbiche D. Validity of asthma diagnoses recorded in the Medical Services database of Quebec. Pharmacoepidemiol Drug Saf. 2006 Apr;15(4):245-52. |
| R14-0353 | Ekström MP, Jogréus C, Ström KE. Comorbidity and sex-related differences in mortality in oxygen-dependent chronic obstructive pulmonary disease. PLoS One. 2012;7(4):e35806. |
| R14-0354 | ENCePP. EU PAS Register. European Network of Centres for Pharmacoepidemiology and Pharmacovigilance; 7 January 2014. Available at: website: encepp_eu/encepp_studies/indexRegister.shtml. Accessed 8 January 2014. |
| R14-0356 | Köster M, Asplund K, Johansson A, Stegmayr B. Refinement of Swedish administrative registers to monitor stroke events on the national level. Neuroepidemiology. 2013;40(4):240-6. |
| R14-0357 | Ludvigsson JF, Andersson E, Ekbom A, Feychting M, Kim JL, Reuterwall C, et al. External review and validation of the Swedish national inpatient register. BMC Public Health. 2011;11:450. |
| R14-0359 | Thomsen RW, Lange P, Hellquist B, Frausing E, Bartels PD, Krog BR, et al. Validity and underrecording of diagnosis of COPD in the Danish National Patient Registry. Respir Med. 2011 Jul;105(7):1063-8. |
| R14-0443 | NOMESCO. NOMESCO classification of surgical procedures, version 1.16:2012. Copenhagen: Nordic Medico-Statistical Committee; 2011. |

Proprietary confidential information © 2014 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

R14-0444 Socialstyrelsen. The National Patient Register. Swedish National Board of Health and Welfare; 2013. Available at: website: socialstyrelsen.se/register/halsodataregister/patientregistret/inenglis h. Accessed 13 February 2013.

R14-0456 Inghammar M, Engstrom G, Lofdahl CG, Egesten A. Validation of a COPD diagnosis from the Swedish Inpatient Registry. Scand J Public Health. 2012 Dec;40(8):773-6.

#### 13.2 UNPUBLISHED REFERENCES

Not applicable

Proprietary confidential information © 2014 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

### ANNEX 1. LIST OF STAND-ALONE DOCUMENTS

None

Proprietary confidential information © 2014 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

### ANNEX 2. ENCEPP CHECKLIST FOR STUDY PROTOCOLS

Proprietary confidential information © 2014 Boehringer Ingelheim International GmbH or one or more of its affiliated companies





European Network of Centres for Pharmacoepidemiology and Pharmacovigilance

Doc.Ref. EMA/540136/2009

#### **ENCePP Checklist for Study Protocols (Revision 2, amended)**

Adopted by the ENCePP Steering Group on 14/01/2013

The European Network of Centres for Pharmacoepidemiology and Pharmacovigilance (ENCePP) welcomes innovative designs and new methods of research. This Checklist has been developed by ENCePP to stimulate consideration of important principles when designing and writing a pharmacoepidemiological or pharmacovigilance study protocol. The Checklist is intended to promote the quality of such studies, not their uniformity. The user is also referred to the ENCePP Guide on Methodological Standards in Pharmacoepidemiology which reviews and gives direct electronic access to guidance for research in pharmacoepidemiology and pharmacovigilance.

For each question of the Checklist, the investigator should indicate whether or not it has been addressed in the study protocol. If the answer is "Yes", the page number(s) of the protocol where this issue has been discussed should be specified. It is possible that some questions do not apply to a particular study (for example in the case of an innovative study design). In this case, the answer 'N/A' (Not Applicable) can be checked and the "Comments" field included for each section should be used to explain why. The "Comments" field can also be used to elaborate on a "No" answer.

This Checklist should be included as an Annex by marketing authorisation holders when submitting the protocol of a non-interventional post-authorisation safety study (PASS) to a regulatory authority (see the Guidance on the format and content of the protocol of non-interventional post-authorisation safety studies). Note, the Checklist is a supporting document and does not replace the format of the protocol for PASS as recommended in the Guidance and Module VIII of the Good pharmacovigilance practices (GVP).

#### Study title:

Drug Utilisation Study for Olodaterol

#### **Study reference number:**

1222.53

Proprietary confidential information © 2014 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| Section 1: Milestones | Yes | No | N/A | Page<br>Number(s) |
|---|---|---|---|---|
| 1.1 Does the protocol specify timelines for | | | | riumber (5) |
| 1.1.1 Start of data collection <sup>1</sup> | $\boxtimes$ | | | 12 |
| 1.1.2 End of data collection <sup>2</sup> | $\boxtimes$ | | | 12 |
| 1.1.3 Study progress report(s) | | | | 12 |
| 1.1.4 Interim progress report(s) | $\boxtimes$ | | | 12 |
| 1.1.5 Registration in the EU PAS register | | | | 12 |
| 1.1.6 Final report of study results. | $\boxtimes$ | | | 12 |

#### Comments:

Timing of PAS registration has not yet been determined.

| Section 2: Research question | Yes | No | N/A | Page<br>Number(s) |
|---|---|---|---|---|
| 2.1 Does the formulation of the research question and objectives clearly explain: | | | | |
| 2.1.1 Why the study is conducted? (e.g. to address an important public health concern, a risk identified in the risk management plan, an emerging safety issue) | | | | 13 |
| 2.1.2 The objective(s) of the study? | $\boxtimes$ | | | 14 |
| 2.1.3 The target population? (i.e. population or subgroup to whom the study results are intended to be generalised) | $\boxtimes$ | | | 15 |
| 2.1.4 Which formal hypothesis(-es) is (are) to be tested? | | | | |
| 2.1.5 If applicable, that there is no <i>a priori</i> hypothesis? | | | | |

#### Comments:

there is no a priori hypothesis and the objective is to measure the relative frequency of off label use among olodaterol and comparator

| Section 3: Study design | Yes | No | N/A | Page<br>Number(s) |
|---|---|---|---|---|
| 3.1 Is the study design described? (e.g. cohort, case-control, randomised controlled trial, new or alternative design) | | | | 15 |
| 3.2 Does the protocol specify the primary and secondary (if applicable) endpoint(s) to be investigated? | | | | 28 |
| 3.3 Does the protocol describe the measure(s) of effect? (e.g. relative risk, odds ratio, deaths per 1000 person-years, absolute risk, excess risk, incidence rate ratio, hazard ratio, number needed to harm (NNH) per year) | | | $\boxtimes$ | |

#### Comments:

<sup>1</sup> Date from which information on the first study is first recorded in the study dataset or, in the case of secondary use of data, the date from which data extraction starts. 2 Date from which the analytical dataset is completely available.

| Section 4: Source and study populations | Yes | No | N/A | Page<br>Number(s) |
|---|---|---|---|---|
| 4.1 Is the source population described? | | | | 18 |
| <ul> <li>4.2 Is the planned study population defined in terms of:</li> <li>4.2.1 Study time period?</li> <li>4.2.2 Age and sex?</li> <li>4.2.3 Country of origin?</li> <li>4.2.4 Disease/indication?</li> <li>4.2.5 Co-morbidity?</li> <li>4.2.6 Seasonality?</li> </ul> | | | | 18<br>18<br>19<br>18 |
| 4.3 Does the protocol define how the study population will be sampled from the source population? (e.g. event or inclusion/exclusion criteria) | | | | 19 |
| Comments: | | | | |
| Section 5: Exposure definition and measurement | Yes | No | N/A | Page<br>Number(s) |
| 5.1 Does the protocol describe how exposure is defined and measured? (e.g. operational details for defining and categorising exposure) | | | | 19 |
| 5.2 Does the protocol discuss the validity of exposure measurement? (e.g. precision, accuracy, prospective ascertainment, exposure information recorded before the outcome occurred, use of validation sub-study) | | | $\boxtimes$ | |
| 5.3 Is exposure classified according to time windows? (e.g. current user, former user, non-use) | | | $\boxtimes$ | |
| 5.4 Is exposure classified based on biological mechanism of action and taking into account the pharmacokinetics and pharmacodynamics of the drug? | | $\boxtimes$ | | |
| 5.5 Does the protocol specify whether a dose-<br>dependent or duration-dependent response is<br>measured? | | | | |
| Comments: This DUS is limited to characterizing the subjects on and group of interest consists of all new users | d before | e first ( | use; ex | posure |
| Section 6: Endpoint definition and measurement | Yes | No | N/A | Page<br>Number(s) |
| 6.1 Does the protocol describe how the endpoints are defined and measured? | | | | 20 |
| 6.2 Does the protocol discuss the validity of endpoint measurement? (e.g. precision, accuracy, sensitivity, specificity, positive predictive value, prospective or retrospective ascertainment, use of validation sub-study) | $\boxtimes$ | | | 19-22 |

| Comments: | | | | |
|---|---|---|---|---|
| Section 7: Confounders and effect modifiers | Yes | No | N/A | Page<br>Number(s) |
| 7.1 Does the protocol address known confounders?<br>(e.g. collection of data on known confounders, methods of controlling for known confounders) | | | | |
| 7.2 Does the protocol address known effect modifiers?<br>(e.g. collection of data on known effect modifiers, anticipated direction of effect) | | | | |
| Comments: | | | | |
| Confounding and effect modification is not expected to study. | be an is | ssue fo | r this c | lescriptive |
| Section 8: Data sources | Yes | No | N/A | Page<br>Number(s) |
| 8.1 Does the protocol describe the data source(s) used in the study for the ascertainment of: | | | | |
| <b>8.1.1</b> Exposure? (e.g. pharmacy dispensing, general practice prescribing, claims data, self-report, face-to-face interview, etc.) | | | | 19 |
| 8.1.2 Endpoints? (e.g. clinical records, laboratory markers or values, claims data, self-report, patient interview including | | | | 20 |
| scales and questionnaires, vital statistics, etc.) 8.1.3 Covariates? | | | | 23 |
| 8.2 Does the protocol describe the information available from the data source(s) on: | | | | |
| 8.2.1 Exposure? (e.g. date of dispensing, drug quantity, dose, number of days of supply prescription, daily dosage, prescriber) | | | | 19 |
| 8.2.2 Endpoints? (e.g. date of occurrence, multiple event, severity measures related to event) | | | | 20 |
| 8.2.3 Covariates? (e.g. age, sex, clinical and drug use history, co-morbidity, co-medications, life style, etc.) | | | | 23 |
| 8.3 Is a coding system described for: | | | | |
| 8.3.1 Diseases? (e.g. International Classification of Diseases (ICD)-10) | | | | 21-22 |
| 8.3.2 Endpoints? (e.g. Medical Dictionary for Regulatory Activities (MedDRA) for adverse events) | $\boxtimes$ | | | 21-22 |
| 8.3.3 Exposure? (e.g. WHO Drug Dictionary, Anatomical Therapeutic Chemical (ATC)Classification System) | | | | 31 |
| 8.4 Is the linkage method between data sources described? (e.g. based on a unique identifier or other) | $\boxtimes$ | | | 29 |
| Comments: | | | | |
| Section 9: Study size and power | Yes | No | N/A | Page<br>Number(s) |
| 9.1 Is sample size and/or statistical power calculated? | $\boxtimes$ | | | 35 |

| Comments: | | | | |
|---|---|---|---|---|
| Section 10: Analysis plan | Yes | No | N/A | Page<br>Number(s) |
| 10.1 Does the plan include measurement of excess risks? | | | | |
| 10.2 Is the choice of statistical techniques described? | $\boxtimes$ | | | 36 |
| 10.3 Are descriptive analyses included? | $\boxtimes$ | | | 36 |
| 10.4 Are stratified analyses included? | $\boxtimes$ | | | 36 |
| 10.5 Does the plan describe methods for adjusting for confounding? | | | | |
| 10.6 Does the plan describe methods addressing effect modification? | | | | |
| Comments: | | | | |
| Confounding and effect modification are not relevant to | this de | scripti | ve stuc | ly |
| Section 11: Data management and quality control | Yes | No | N/A | Page<br>Number(s) |
| 11.1 Is information provided on the management of missing data? | $\boxtimes$ | | | 35 |
| 11.2 Does the protocol provide information on data storage? (e.g. software and IT environment, database maintenance and anti-fraud protection, archiving) | | | | 38 |
| 11.3 Are methods of quality assurance described? | $\boxtimes$ | | | 38 |
| 11.4 Does the protocol describe possible quality issues related to the data source(s)? | | $\boxtimes$ | | |
| 11.5 Is there a system in place for independent review of study results? | | | | |
| Comments: 11.1-11.3 This is a core protocol that will be implement institution that are qualified and have available staffing i.e. after EMA review, olodaterol is launched. At that tir management for each data source and corresponding requality control and data security, can be specified. 11. 5 To date no advisory board is planned. | at the me the | time of<br>specifi | f study<br>cs of d | initiation,<br>ata |
| Section 12: Limitations | Yes | No | N/A | Page<br>Number(s) |
| 12.1 Does the protocol discuss: 12.1.1 Selection biases? 12.1.2 Information biases? (e.g. anticipated direction and magnitude of such biases, | | | | 37-38 |
| (2.3. a.m. para and and magnitude of odd) bladed | | шШ | | 37 30 |

| Section 12: Limitations | Yes | No | N/A | Page<br>Number(s) |
|---|---|---|---|---|
| validation sub-study, use of validation and external data, analytical methods) | | _ | | |
| 12.2 Does the protocol discuss study feasibility? (e.g. sample size, anticipated exposure, duration of follow-up in a cohort study, patient recruitment) | | | | 37-38 |
| 12.3 Does the protocol address other limitations? | $\boxtimes$ | | | 37-38 |
| Comments: | | | | |
| Section 13: Ethical issues | Yes | No | N/A | Page<br>Number(s) |
| 13.1 Have requirements of Ethics<br>Committee/Institutional Review Board approval<br>been described? | | | | 40 |
| 13.2 Has any outcome of an ethical review procedure been addressed? | | $\boxtimes$ | | |
| 13.3 Have data protection requirements been described? | | $\boxtimes$ | | 35 |
| Comments: | <b>'</b> | | l | |
| For this core protocol, the data protection procedures procedures and more details will be added into data s | | | | |
| Section 14: Amendments and deviations | Yes | No | N/A | Page |
| Section 14: Amendments and deviations | Yes | No | N/A | Page<br>Number(s) |
| Section 14: Amendments and deviations 14.1 Does the protocol include a section to document future amendments and deviations? | | No | N/A | _ |
| 14.1 Does the protocol include a section to document | | No | N/A | Number(s) |
| 14.1 Does the protocol include a section to document future amendments and deviations? | | No | N/A | Number(s) |
| 14.1 Does the protocol include a section to document future amendments and deviations? | | No | N/A | Number(s) |
| 14.1 Does the protocol include a section to document future amendments and deviations? Comments: Section 15: Plans for communication of study | | | | Number(s) 11 Page |
| 14.1 Does the protocol include a section to document future amendments and deviations? Comments: Section 15: Plans for communication of study results 15.1 Are plans described for communicating study | Yes | | | Number(s) 11 Page Number(s) |
| 14.1 Does the protocol include a section to document future amendments and deviations? Comments: Section 15: Plans for communication of study results 15.1 Are plans described for communicating study results (e.g. to regulatory authorities)? 15.2 Are plans described for disseminating study | Yes | | | Page<br>Number(s) |
| 14.1 Does the protocol include a section to document future amendments and deviations? Comments: Section 15: Plans for communication of study results 15.1 Are plans described for communicating study results (e.g. to regulatory authorities)? 15.2 Are plans described for disseminating study results externally, including publication? | Yes | | | Page<br>Number(s) |
| 14.1 Does the protocol include a section to document future amendments and deviations? Comments: Section 15: Plans for communication of study results 15.1 Are plans described for communicating study results (e.g. to regulatory authorities)? 15.2 Are plans described for disseminating study results externally, including publication? Comments: | Yes | | | Page<br>Number(s) |

# ANNEX 3. EVALUATION OF COPD SEVERITY IN AUTOMATED HEALTH DATABASES

Annex Table 3:1 Published definitions of COPD severity in studies conducted in automated health databases

| Reference, Severity | | COPD Seven | rity |
|---|---|---|---|
| Criteria | Mild | Moderate | Severe |
| Integrated Primary Ca | re Information Pro | ject, Netherlands [ <u>P1</u> | 1-13226] |
| With spirometry data, used GOLD criteria [P13-02399] Without spirometry, used methods of Curkendall et al., [R09-0579] Eisner et al., [R13-1392] and Soriano et al. [R08-1492] | At initial COPD symptoms | At least 2 prescriptions of bronchodilators of the same drug class with a maximum interval of 6 months in 1 year | <ul> <li>Severe:</li> <li>Hospitalisation for COPD, or</li> <li>Third course of antibiotics for respiratory infection in 1 year, or</li> <li>Second course of systemic corticosteroids for COPD exacerbation in 1 year</li> <li>Very severe:</li> <li>Oxygen therapy, or</li> <li>Scheduled for lung transplant</li> </ul> |
| Saskatchewan Health, | Canada [R09-0579] | | |
| Case-control study to find severity marker variables, using: • Pre-existing chronic conditions • Recent acute conditions • Recent high use of bronchodilators Specific components of the above are detailed in the article's appendix | Patients ranked into 5 quintiles by likelihood of COPD hospitalisation, from conditional logistic regression model | | Factors in previous 180 days associated with severe COPD: Emphysema Recent nebuliser use Home oxygen therapy Corticosteroid use Frequent bronchodilator use Pneumonia Previous COPD exacerbation |

Proprietary confidential information © 2014 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## Annex Table 3:1 (con't) Published definitions of COPD severity in studies conducted in automated health databases

| *************************************** | | | |
|---|---|---|---|
| , | COPD Severity | | |
| criteria | Mild | Moderate | Severe |
| General Practice Research Database, United Kingdom Soriano [R08-1492] | | | |
| Severity based only on drug data | At first diagnosis of COPD | At least 2 prescriptions of the same COPD drug within 6 months, using data on inhaled or oral bronchodilators, xanthines, cromones, steroids, or combinations | <ul><li>Oxygen therapy, or</li><li>Nebuliser therapy</li></ul> |

COPD = Chronic Obstructive Pulmonary Disease; GOLD = Global Initiative for Chronic Obstructive Lung Disease.

<sup>1</sup> This database is now known as Clinical Practice Research Datalink.

# ANNEX 4. CODES FOR COMORBIDITIES AND OTHER MEDICATIONS

Annex Table 4:1 Other comorbidity

| Disease Description | ICD-10 Code | ICD-9 Code |
|---|---|---|
| Cardiovascular diseases | 100-199 | 390-459 |
| Ischaemic heart disease | I20-I25 or coronary reperfusion surgery and procedures | 410-414 or coronary reperfusion surgery and procedures |
| Angina pectoris | I20 | 413, 411.1 |
| Acute myocardial infarction | I21 | 410 |
| Other acute or subacute ischaemic heart disease | 122-124 | 411.0, 411.8 |
| Chronic ischaemic heart disease | I25 | 412, 414 |
| Coronary reperfusion surgery and procedures | List of codes to be<br>developed according to<br>each database dictionary | List of codes to be<br>developed according to<br>each database dictionary |
| Arrhythmias | I47-I49 | 427.0-427.4, 427.6-427.9 |
| Paroxysmal tachycardia | I47 | 427.0-427.2 |
| Ventricular tachycardia | I47.0, I47.2 | 427.1 |
| Supraventricular tachycardia and unspecified | I47.1, I47.9 | 427.0, 427.2 |
| Atrial fibrillation and flutter | I48 | 427.3 |
| Other cardiac arrhythmias | I49 | 427.4, 427.6, 427.8, 427.9 |
| Ventricular fibrillation and flutter | 149.0 | 427.4 |
| Other cardiac arrhythmias | I49.1-I49.9 | 427.6, 427.8, 427.9 |
| Conduction disorders | I44-I45 | 426 |
| Cardiac arrest | I46 | 427.5 |
| Heart failure | I50 | 428 |
| Cerebrovascular disease | I60-I69, G45 | 430-438 |
| Cerebral haemorrhage (subarachnoid, intracerebral, other non-traumatic) | 160-162 | 430-432 |

Annex Table 4:1 (con't) Other comorbidity

| <b>Disease Description</b> | ICD-10 Code | ICD-9 Code |
|---|---|---|
| Cardiovascular diseases | 100-199 | 390-459 |
| Cerebral infarction and stroke | I63, I64, G46.5 | 433.1, 434.1, 436 |
| Transient ischaemic attack | G45 | 435 |
| Other cerebrovascular disease and sequelae of cerebrovascular disease | I65-I69 | 433.0, 434.0, 437, 438 |
| Hypertension and hypertensive heart disease | 110-115 | 401-405 |
| Diseases of arteries, arterioles, and capillaries | I70-I79, and peripheral arterial revascularisation procedures | 440-449 and peripheral arterial revascularisation procedures |
| Peripheral arterial revascularisation procedures | List of codes to be<br>developed according to<br>each database dictionary | List of codes to be<br>developed according to<br>each database dictionary |
| Other form of heart diseases | 100-109, 130-143, 180-199 | 390-398, 420-425, 429,<br>440-459 |
| Hyperlipidaemia | E78 | 272 |
| Diabetes mellitus | E10-E14 | 250 |
| Renal disease | N00-N39 | 580-599 |
| Chronic kidney disease | N18 | 585 |
| Other renal disorders | N00-N17, N19, N25-N39 | |
| Anaemias | D50-D64 | 280-285 |
| Nutritional anaemias | D50-D53 | 280-281 |
| Iron deficiency anaemias | D50 | 280 |
| Other anaemias | D55-D64 | 282-285 |
| Peptic ulcer disease | K25-K28 | 531-534 |
| Liver disease | K70-K77 | 570-573 |
| Osteoporosis | M80-M82 | 733.0 |
| Rheumatoid arthritis and other inflammatory arthropathies | M05-M14 | 712-714, 716, 696.0 |
| Systemic connective tissue diseases | M30-M36 | 710 |
| Malignancy | C00-C97 | 140-209 |
| Depressive disorders | F32-F33 | 311, |
| Pregnancy (at the index date) | O00-O48 | 630-649 |

ICD-10 = International Statistical Classification of Diseases and Related Health Problems, 10th Revision; ICD-9 = International Classification of Diseases, 9th Revision.

Annex Table 4:2 Anatomical Therapeutic Chemical codes for comedications

| Medication Description | ATC Code |
|-----------------------------|----------|
| Respiratory medications | |
| Inhaled SAMAs | |
| Ipratropium bromide | R03BB01 |
| Oxitropium bromide | R03BB02 |
| Inhaled LAMAs | |
| Tiotropium bromide | R03BB04 |
| Aclidinium bromide | R03BB05 |
| Glycopyrronium bromide | R03BB06 |
| Inhaled SABAs | |
| Salbutamol | R03AC02 |
| Terbutaline | R03AC03 |
| Fenoterol | R03AC04 |
| Rimiterol | R03AC05 |
| Hexoprenaline | R03AC06 |
| Isoetarine | R03AC07 |
| Pirbuterol | R03AC08 |
| Tretoquinol | R03AC09 |
| Carbuterol | R03AC10 |
| Tulobuterol | R03AC11 |
| Clenbuterol | R03AC14 |
| Reproterol | R03AC15 |
| Procaterol | R03AC16 |
| Bitolterol | R03AC17 |
| Indacaterol | R03AC18 |
| Inhaled LABAs | |
| Salmeterol | R03AC12 |
| Formoterol | R03AC13 |
| Inhaled glucocorticosteroid | |
| Beclometasone | R03BA01 |
| Budesonide | R03BA02 |

Annex Table 4:2 (con't) Anatomical Therapeutic Chemical codes for comedications

| Medication Description | ATC Code |
|---|---|
| Respiratory medications | |
| Flunisolide | R03BA03 |
| Betamethasone | R03BA04 |
| Fluticasone | R03BA05 |
| Triamcinolone | R03BA06 |
| Mometasone | R03BA07 |
| Ciclesonide | R03BA08 |
| Fixed combinations of SABAs and SAMAs | ATC codes not available <sup>1</sup> |
| Fixed combinations of SABAs and ICSs | ATC codes not available <sup>1</sup> |
| Fixed combinations of LABAs and ICSs | ATC codes not available <sup>1</sup> |
| Systemic glucocorticosteroids | H02AB |
| Systemic beta2-agonists | R03CC |
| Xanthines and adrenergics | R03DA, R03DB |
| Roflumilast | R03DX07 |
| Nasal glucocorticosteroids | R01AD |
| Omalizumab | R03DX05 |
| Leukotriene receptor antagonists | R03DC |
| Cromoglicic acid | R03BC01 |
| Nedocromil | R03BC03 |
| Methotrexate | L04AX03 |
| Ciclosporin | L04AD01 |
| Gold preparations | M01CB |
| Oxygen therapy | V03AN01 |
| Nebuliser therapy | ATC codes not available <sup>1</sup> |
| Cardiovascular medications | All codes listed below in section<br>Cardiovascular medications |
| Cardiac glycosides and antiarrhythmics, Classes I and III | C01A, C01B |
| Vasodilators used in cardiac diseases | C01D |
| Other cardiac preparations | C01B, C01C |
| Diuretics | C03 |
| Peripheral vasodilators | C04 |

Annex Table 4:2 (con't) Anatomical Therapeutic Chemical codes for comedications

| Annex Table 4:2 (con't) Anatomical Therapeutic Chemical codes for comedications | |
|---|---|
| Medication Description | ATC Code |
| Cardiovascular medications | All codes listed below in section<br>Cardiovascular medications |
| Beta blocking agents | C07 |
| Calcium channel blockers | C08 |
| Antihypertensives | C02 |
| Agents acting on the renin-angiotensin system | C09 |
| Angiotensin-converting-enzyme inhibitors | C09A, C09B |
| Angiotensin II receptor antagonists | C09C, C09D |
| Renin-inhibitors | C09X |
| Lipid-modifying agents | C10 |
| HMG CoA reductase inhibitors (statins) | C10AA |
| Other lipid-modifying agents | C10AB, C10AC, C10AD, C10AX |
| HMG CoA reductase inhibitors (statins), other combination | C10BX |
| Antithrombotic agents | B01 |
| Platelet aggregation inhibitors | B01AC |
| Systemic antibacterials | J01 |
| Iron preparations | B03A |
| Proton pump inhibitors | A02BC |
| Drugs used in diabetes | A10 |
| Insulins | A10A |
| Blood glucose-lowering drugs | A10B, A10X |
| Drugs for musculoskeletal system | M01A, N02BA, M01B, M01C |
| Antiinflammatory and antirheumatic products, non-steroids (nonsteroidal anti-inflammatory drugs) | M01A |
| Acetylsalicylic acid (other analgesics and antipyretics) | N02BA |
| Other antirheumatic agents:<br>Antiinflammatory/antirheumatic agents in<br>combination, specific antirheumatic agents | M01B-M01C |
| Antidepressants | N06A |
| Selective serotonin reuptake inhibitors | N06AB |
| Antineoplastic agents | L01 |

**BI Study Number 1222.53** 

c02329987-02

Proprietary confidential information © 2014 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Annex Table 4:2 (con't) Anatomical Therapeutic Chemical codes for comedications

| <b>Medication Description</b> | ATC Code |
|---|---|
| Immunosuppressants | L04 |
| Antivirals for systemic use | J05 |
| Hormone-replacement therapy: Estrogens, progestogensprogestogens, and estrogens in combination | G03C, G03D, G03F |
| Drugs used in nicotine dependence | N07BA |

ATC = Anatomical Therapeutic Chemical; ICS = Inhaled Glucocorticosteroid; LABA = Long-Acting Beta2-Agonist; LAMA = Long-Acting Muscarinic Antagonist; SABA = Short-Acting Beta2-Agonist; SAMA = Short-Acting Muscarinic Antagonist.

<sup>1</sup> The national drug code of each database country will be used to identify medications without an individual ATC code. Source: WHO Collaborating Centre for Drug Statistics Methodology. ATC/DDD Index 2013. Updated 20 December 2012. Available at: website: whocc.no/atc\_ddd\_index/. Accessed 21 January 2013.

**BI Study Number 1222.53** 

Proprietary confidential information © 2014 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## ANNEX 5. DETAILS ON EACH DATABASE FROM THE FEASIBILITY REPORT (1 NOVEMBER 2013)

#### PHARMO, THE NETHERLANDS

#### **Database Characteristics**

#### **Database Description**

The PHARMO Database Network consists of multiple databases containing data files on approximately 3.2 million community-dwelling inhabitants in geographically defined areas covering approximately 20% of the Netherlands. Annex Figure 5:1 shows the databases included in the PHARMO Database Network. Data sources include information from GPs, community pharmacies, hospitals, and laboratory sources.



GP = General Practitioner; PRO = Patient-Reported Outcome.

#### Annex Figure 5:1 Data sources within the PHARMO Database Network

The patients covered in each database are not necessarily included in all of the databases, as some of the geographical areas overlap partially; but if patients are in more than one database, they can be linked to construct the medical history as shown in Annex Figure 5:2 Thus, high-quality research has been conducted with ascertainment of patient demographics, drug dispensings, hospital morbidity, clinical laboratory results, and date of death.



GP = general practitioner.

Annex Figure 5:2 Schematic overview of overlap example among databases included in the PHARMO Database Network